CLINICAL TRIAL: NCT02382822
Title: Copenhagen Comorbidity in HIV Infection Study
Acronym: COCOMO
Status: Active, not recruiting | Type: Observational
Sponsor: Susanne Dam Nielsen, MD, DMSc (Other)
Responsible Party: Sponsor-Investigator, Susanne Dam Nielsen, MD, DMSc, Professor, MD, DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-8-2014-004
Record Dates: First submitted 2015-03-03; First posted 2015-03-09 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: HIV; COPD; CVD; Liver Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Routine biochemistry, whole blood, plasma, peripheral blood mononuclear cells (PBMCs), DNA and RNA from buffy coat, plasma, and red blood cells (RBC).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- HIV infected: Exposure to: Computed tomography(CT) of chest and upper abdomen, CT angiography(CTa) of heart, spirometry, mouth wash, eNO assessment, ankle brachial pressure index, fibroscan, blood sampling
  Interventions: Other: No intervention.
- HIV uninfected: Exposure to: Computed tomography(CT) of chest and upper abdomen, CT angiography(CTa) of heart, spirometry, eNO assessment, ankle brachial pressure index, blood sampling
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention.

SUMMARY:
Despite efficient antiretroviral treatment for HIV infection, decrease in life expectancy remains. Excess mortality is mainly due to non-AIDS co-morbidity including cardiovascular, pulmonary, and liver related diseases. Both HIV-unrelated and HIV-related risk factors probably contribute to this pattern. At present, most evidence regarding co-morbidity in HIV infection rely on cross-study comparisons of HIV-infected persons with published population rates and few prospective studies in U.S. cohorts. Using well characterized participants from the Copenhagen General Population Study (CGPS) as controls, we aim to include >1500 HIV-infected persons in the COCOMO study to determine if co-morbidity is more prevalent or develops at a higher rate in HIV-infected persons. The study will asses 1) cardiovascular, 2) pulmonary and 3) liver-related co-morbidity using uniformly collected data in the two cohorts. The investigators aim to study the relative impact of HIV-unrelated and HIV-related factors on development of co-morbidity.

DETAILED DESCRIPTION:
Primary hypothesis:

Cardiovascular disease:

- HIV infection is independently associated with higher prevalence of coronary atherosclerosis (assessed by CT angiography)

Obstructive pulmonary disease:

- HIV infection is independently associated with higher prevalence of COPD, and independently associated with loss of lung function

Liver disease:

- HIV infection is independently associated with liver steatosis, steatohepatitis and liver fibrosis

Lipid and fat metabolism:

- HIV infection is independently associated with alterations in adipose fat tissue and dyslipidemia

Secondary hypothesis:

Cardiovascular disease:

* Viral load and CD4 are independently associated with coronary atherosclerosis (assessed by CT angiography) in HIV-infected individuals.
* Levels of inflammatory markers can predict coronary atherosclerosis in HIV-infected individuals.
* Microbial translocation and metabolism are associated with coronary atherosclerosis in HIV-infected individuals.
* Endothelial dysfunction (assessed by arterial elastography) can predict coronary atherosclerosis in HIV-infected individuals

Obstructive pulmonary disease:

* Viral load and CD4 is independently associated with emphysema
* HIV is independently associated with pulmonary hypertension (assessed by CT angiography), and obstructive lung disease is independently associated with airway obstruction
* PCP colonization in HIV infected patients is independently associated with obstructive lung disease, emphysema and loss of lung function.
* Inflammatory markers in HIV infected patients are associated with obstructive lung disease and loss of lung function

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* HIV infected
* aged 20-100 years

Exclusion Criteria:

* patients that are unable to understand information material

Computed tomography (CT):

* contraindications to CT and contrast (i.e. pregnancy, renal impairment, allergy to contrast media, allergy or contraindication to beta blocking agent, body weight more than 120kg, evidence of ongoing myocardial ischemia, heart rhythm precluding EKG gating)

Spirometry:

* relative contraindications to spirometry (i.e. chest, abdominal or eye surgery within the 3 months before baseline spirometry, and known retinal detachment)
* allergy or contraindications to salbutamol (i.e. >110 bpm, or a known uncontrolled cardiac condition (i.e. unstable coronary artery disease, decompensated heart failure)
* a respiratory illness with at least two symptoms of breathlessness, cough, wheezing, or increase in sputum production within 6 weeks.

MRI:

* Implants (e.g. pacemaker, coclea implants, insulin pumps)
* Claustrophobia
* Pregnancy

Liver Biopsy:

* Risk of bleeding
* Infection in puncture site

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected patients.
Sampling Method: Non-Probability Sample
Enrollment: 1099 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Coronary atherosclerosis | Baseline cross-sectional data and after 2 years follow-up
  Prevalence of coronary atherosclerosis; electrocardiographic abnormalities and peripheral artery disease
Obstructive pulmonary disease | Baseline cross-sectional data and after 2 years follow-up
  Emphysema, airflow limitation,
Liver disease | Baseline cross-sectional data and after 2 years follow-up
  Prevalence of hepatic steatosis, steatohepatitis and liver fibrosis
Lipid and fat metabolism | Baseline cross-sectional data and after 2 years follow-up
  Visceral adipose tissue, dyslipidemia, gut microbiota
Inflammation and clonal hematopoiesis | Baseline cross-sectional data and after 2 years follow-up
  Cytokines (e.g. IL-6, TNF-alfa), cell subsets (e.g. Tregs, Th17)

SECONDARY OUTCOMES:
Emphysema, P. jirovecii colonization | Baseline data(cross-sectional data)
  Secondary pulmonary outcome measures
Depression | Baseline data (cross-sectional data)
  Major Depression Inventory Score, kynurenin/tryptophan ratio
Bone metabolism | Baseline data(cross-sectional data) assessed after two years
  Bone mineral density
Hematological abnormalities | Baseline data(cross-sectional data)
  Anemia, trombocytopenia, leukopenia
Renal function | Baseline data(cross-sectional data)
  Kidney function

CONTACTS AND LOCATIONS:
Overall Officials: Susanne D Nielsen, Professor, MD, DMSc, Principal Investigator — Department of Infectious Diseases, Copenhagen University Hospital - Rigshospitalet; Thomas L Benfield, Professor, MD, DMSc, Study Director — Department of Infectious Diseases, Copenhagen University Hospital - Amager and Hvidovre; Klaus F Kofoed, Professor, MD, PhD, DMSc, Study Director — Department of Cardiology, Copenhagen University Hospital - Rigshospitalet; Lars V Køber, Professor, MD, PhD, DMSc, Study Director — Department of Cardiology, Copenhagen University Hospital - Rigshospitalet; Børge G Nordestgaard, Professor, MD, DMSc, Study Director — Department of Clinical Biochemistry, Copenhagen University Hospital - Herlev and Gentofte; Shoaib Afzal, Professor, MD, DMSc, Study Director — Department of Clinical Biochemistry, Copenhagen University Hospital - Herlev and Gentofte
Locations (2):
- Denmark (2):
  - Copenhagen University Hospital - Rigshospitalet, Copenhagen
  - Copenhagen University Hospital - Amager and Hvidovre, Hvidovre

REFERENCES:
- [Derived] Thudium RF, Ringheim H, Ronit A, Hoel H, Benfield T, Mocroft A, Gerstoft J, Troseid M, Borges AH, Ostrowski SR, Vestbo J, Nielsen SD. Independent Associations of Tumor Necrosis Factor-Alpha and Interleukin-1 Beta With Radiographic Emphysema in People Living With HIV. Front Immunol. 2021 Apr 14;12:668113. doi: 10.3389/fimmu.2021.668113. eCollection 2021. PMID 33936110
- [Derived] Kirkegaard-Klitbo DM, Thomsen MT, Gelpi M, Bendtsen F, Nielsen SD, Benfield T. Hepatic Steatosis Associated With Exposure to Elvitegravir and Raltegravir. Clin Infect Dis. 2021 Aug 2;73(3):e811-e814. doi: 10.1093/cid/ciab057. PMID 33493297
- [Derived] Ronit A, Lundgren J, Afzal S, Benfield T, Roen A, Mocroft A, Gerstoft J, Nordestgaard BG, Vestbo J, Nielsen SD; Copenhagen Co-morbidity in HIV infection (COCOMO) study group. Airflow limitation in people living with HIV and matched uninfected controls. Thorax. 2018 May;73(5):431-438. doi: 10.1136/thoraxjnl-2017-211079. Epub 2018 Jan 13. PMID 29331988
- [Derived] Ronit A, Kristensen T, Klitbo DM, Gelpi M, Kalhauge A, Benfield T, Gerstoft J, Lundgren J, Vestbo J, Kofoed KF, Nielsen SD. Incidental lung cancers and positive computed tomography images in people living with HIV. AIDS. 2017 Sep 10;31(14):1973-1977. doi: 10.1097/QAD.0000000000001600. PMID 28857778
- [Derived] Ronit A, Mathiesen IH, Gelpi M, Benfield T, Gerstoft J, Pressler T, Christiansen A, Lundgren J, Vestbo J, Dam Nielsen S. Small airway dysfunction in well-treated never-smoking HIV-infected individuals. Eur Respir J. 2017 Mar 2;49(3):1602186. doi: 10.1183/13993003.02186-2016. Print 2017 Mar. No abstract available. PMID 28254767
- [Derived] Ronit A, Haissman J, Kirkegaard-Klitbo DM, Kristensen TS, Lebech AM, Benfield T, Gerstoft J, Ullum H, Kober L, Kjaer A, Kofoed K, Vestbo J, Nordestgaard B, Lundgren J, Nielsen SD. Copenhagen comorbidity in HIV infection (COCOMO) study: a study protocol for a longitudinal, non-interventional assessment of non-AIDS comorbidity in HIV infection in Denmark. BMC Infect Dis. 2016 Nov 26;16(1):713. doi: 10.1186/s12879-016-2026-9. PMID 27887644